CLINICAL TRIAL: NCT00796081
Title: Open-label Study to Evaluate the Safety and Pharmacokinetics of Single- and Multiple-dose Extended-release OROS Paliperidone in Pediatric Subjects (=10 to =17 Years of Age) With Schizophrenia, Schizoaffective Disorder, or Schizophreniform Disorder
Brief Title: A Safety and Pharmacokinetic Study of ER OROS Paliperidone in Pediatric Patients With Schizophrenia, Schizoaffective Disorder, or Schizophreniform Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002371
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders
Keywords: Schizophrenia; Schizoaffective disorder; Schizophreniform disorders; Mood disorders; Antipshychotic drugs; Pediatrics; ER OROS Paliperidone, Paliperidone ER
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: ER OROS paliperidone, paliperidone ER

SUMMARY:
The purposes of this study are to characterize the pharmacokinetics of paliperidone after single- and multiple-dose administration of paliperidone ER in children and adolescent patients (>= 10 to <= 17 years of age) with schizophrenia, schizoaffective disorder, or schizophreniform disorder and to evaluate the safety and tolerability of paliperidone ER in this patient population.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, open-label, multiple-dose study in children and adolescent patients >= 10 to <= 17 years of age with schizophrenia, schizoaffective disorder, or schizophreniform disorder. The study includes 3 dosage groups (0.086, 0.129, and 0.171 mg/kg/day paliperidone ER), which will be studied in a sequential ascending design, so that the safety of the drug can be properly evaluated with a lower dosage before proceeding to the next higher dosage. The 3 dosages are approximately 6, 9, and 12 mg/day in adults. Within each dosage group, patients will be randomly assigned to 1 of 2 pharmacokinetic sampling schedules in a 1:1 ratio. For each dosage group, the study consists of a screening phase (for a maximum of 21 days); a 2-day, single-dose pharmacokinetic and tolerability evaluation phase; a 7-day multiple-dose phase, with evaluation of pharmacokinetics and tolerability; and an end-of-study visit. Following the completion of all patients in a given dosage group, the sponsor will evaluate the safety and tolerability of the treatment, in order to determine whether to proceed to the next higher or lower dosage level. The first group will start at 0.086 mg/kg/day. The hypothesis is that paliperidone ER will be well tolerated in children and adolescent patients with schizophrenia, schizoaffective disorder, or schizophreniform disorder, and will display the expected pharmacokinetic characteristics in this population. Paliperidone ER 0.086, 0.129, and 0.171 mg/kg/day, oral administration, single dose on Day 1 of study followed by once daily dosing on Days 3 to 9.

ELIGIBILITY:
Inclusion Criteria:

* Patients' height and weight must be within the 5th to 95th Physical Growth National Center for Health Statistics percentiles for age and sex
* Patients must have a diagnosis of schizophrenia of any subtype (295.10
* 295.20
* 295.30
* 295.60
* 295.90), schizoaffective disorder (295.70), or schizophreniform disorder (295.40), according to the DSM-IV-TR
* Patients must be healthy (other than the DSM-IV-TR classification), on the basis of the screening medical history, physical examination, 12-lead ECG, and clinical laboratory tests (hematology, serum chemistry, and urinalysis). Patients with laboratory results outside the normal reference range can be included only if the investigator, upon consultation with the sponsor, judges the deviations as not clinically significant
* QT values must be within normal limits and patients must have a CGI-S score of less than or equal to 3
* Female patients must be premenarchal, surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) for at least 1 month before study entry and throughout the study, have a negative serum beta-human chorionic gonadotropin pregnancy test at screening, and a negative urine pregnancy test on Day 1
* Patients must sign an informed assent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study, with Parent(s) or the legal guardian(s) of each patient signing an informed consent document indicating that they understand the purpose of and the procedures required for the study and give permission for their child's participation in the study and a responsible person must be available to accompany the patient to the investigational site at each visit
* Patients must agree to be hospitalized at any time during the study, and their parent(s) or legal guardian(s) must consent, if it is deemed clinically necessary by the investigator.

Exclusion Criteria:

* Patients with an active DSM-IV-TR axis I diagnosis other than schizophrenia, schizoaffective disorder, or schizophreniform disorder
* Patients with a history of DSM-IV-TR diagnosis of substance dependence within 6 months before screening (nicotine and caffeine dependence are not exclusionary) or patients who are involuntarily committed to psychiatric hospitalization
* Patients with a significant risk of suicidal or violent ideation or behavior, as judged by the clinical investigator
* Female patients who are pregnant, who plan to become pregnant during the study, or who are breast-feeding
* Patients with any medical condition that can potentially alter the absorption, metabolism, or excretion of the study drug (e.g., Crohn's disease, severe gastrointestinal narrowing [pathologic or iatrogenic], liver disease, or renal disease)
* Patients with a history of any malignancy, with the exception of basal cell carcinoma, in the past 5 years
* Patients with a history of a positive result for any serology test (e.g., human immunodeficiency virus, hepatitis), with a history of neuroleptic malignant syndrome

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2006-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
to characterize the pharmacokinetics of paliperidone after single- and multiple-dose oral administrations of paliperidone ER in children and adolescent patients (>= 10 to <= 17 years of age)

SECONDARY OUTCOMES:
to evaluate the safety and tolerability of paliperidone ER in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A safety and pharmacokinetic study of ER OROS paliperidone in pediatric patients with schizophrenia, schizoaffective disorder, or schizophreniform disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=473&filename=CR002371_CSR.pdf